CLINICAL TRIAL: NCT03845933
Title: Comparing Right Colon Adenoma and Hyperplastic Polyp Miss Rate in Colonoscopy Using Water Exchange and Carbon Dioxide Insufflation: A Prospective Randomized Controlled Trial
Brief Title: Right Colon Polyp Miss Rates of Water Exchange and Carbon Dioxide Insufflation Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Responsible Party: Principal Investigator, Chi-Liang Cheng, M.D., Evergreen General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGH-2019
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Right Colon Adenoma Miss Rate; Right Colon Hyperplastic Polyp Miss Rate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The second endoscopist will perform tandem right colon examination and is blinded to the insertion method used by the first endoscopist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water exchange (WE) colonoscopy (Active Comparator): Water exchange will be used during colonoscopy insertion. Upon arriving at the cecum, CO2 will be opened. The scope will be withdrawn to the hepatic flexure. All polyps identified will be resected (colon polypectomy). The scope will be reinserted into the cecum by the first endoscopist. A tandem inspection of right colon will be performed by a second endoscopist. All polyps found herein will be counted as the missed polyps. After the second withdrawal to the distal hepatic flexure, the remainder of the colon will be examined in a standard manner by the first endoscopist.
  Interventions: Procedure: Colon polypectomy
- CO2 insufflation colonoscopy (Active Comparator): The colonoscopy is performed in the usual fashion, with minimal insufflation required to aid insertion. Cleaning will be performed entirely during withdrawal. Upon arriving at the cecum, CO2 insufflation will be used and the scope will be withdrawn to the hepatic flexure. All polyps identified will be resected (colon polypectomy). Then the scope will be reinserted into the cecum by the first endoscopist using CO2. A tandem inspection of the right colon will then be performed by a second endoscopist. All polyps found herein will be counted as the missed polyps. After the second withdrawal to the mark of distal hepatic flexure, the remainder of the colon will be examined in a standard manner by the first endoscopist.
  Interventions: Procedure: Colon polypectomy

INTERVENTIONS:
Procedure: Colon polypectomy — Polyp search and resection will be performed during the withdrawal phase in both groups. Insertion polypectomy will not be performed. All proximal colon polyps will be removed irrespective of their size and appearance.

SUMMARY:
This will be a prospective randomized controlled trial comparing CO2 insufflation and WE in terms of right colon combined adenoma miss rate (AMR) and hyperplastic polyp miss rate (HPMR) by tandem inspection. It will be a single-site study conducted in Taiwan.

DETAILED DESCRIPTION:
This will be a prospective RCT comparing CO2 insufflation and WE in terms of right colon combined AMR and HPMR by tandem inspection. It is originally designed as a multicenter study conducted in three community hospitals in Taiwan. Consecutive patients will be enrolled from April 2019 to October 2020. A written informed consent will be obtained from all participating patients. The study has obtained ethical approval from the Joint Institutional Review Board of Taiwan (19-002-T-1) and has been registered with ClinicalTrials.gov (NCT03845933). Due to delay in obtaining IRB approval in two of the participating hospitals (Dalin Tzu-Chi Hospital obtained IRB approval in late May 2019 and has not recruited any patient; Taipei Medical University Hospital has not obtained IRB approval in early June 2019) and rapid recruitment of Evergreen General Hospital since April 2019, which has recruited and completed more than 90 patients in the end of May 2019, we have amended the study design from multicenter study to single-center study and have obtained the approval of this amendment from the Joint Institutional Review Board of Taiwan. Consecutive patients aged 45 years or older undergoing colonoscopy for screening, surveillance, and positive FIT will be considered for enrollment from April 2019 to October 2020. Participants will be randomized in a 1:1 ratio to undergo either the CO2 insufflation colonoscopy (CO2 group) or WE colonoscopy (WE group). Colonoscopies will be performed by two board-certified colonoscopists (Chi-Liang Cheng, Yen-Lin Kuo). Standard colonoscopes (CF-Q260AL/I; Olympus Medical Systems Corp., Tokyo, Japan) will be used. All colonoscopists have performed more than 1000 conventional colonoscopies. Hands-on coaching by a WE expert (Felix W. Leung) to standardize the WE method has been completed. Each colonoscopist has completed 100 cases of WE learning curve. Felix W. Leung will be involved in the study design, data analyses, and report preparation, but not in patient enrollment. CO2 insufflation will be used for CO2 group and the withdrawal phase of the WE group. In the WE group, the air pump will be turned off before starting the procedure. During the insertion phase, air and residual water or feces in the rectum will be aspirated, and then the colon will be irrigated with warm water. When the cecum is reached, CO2 will be opened. In the CO2 group, colonoscopy is performed in the usual fashion, with minimal insufflation required to aid insertion. Cleaning in the CO2 group will be performed entirely during withdrawal. Upon arriving at the cecum, CO2 insufflation will be used in both groups and the scope will be withdrawn from the cecum to the hepatic flexure, with inspection of the mucosa at the same time. All polyps identified will be resected and sent for pathology evaluation. The most distal part of the hepatic flexure will be marked by a forceps biopsy and then the scope will be reinserted into the cecum by the first endoscopist using CO2 insufflation. A tandem inspection of the right colon will then be performed by a second endoscopist blinded to the insertion method in both study groups. All polyps found herein will be counted as the missed polyps. After the second withdrawal to the mark of distal hepatic flexure, the remainder of the colon will be examined in a standard manner by the first endoscopist. Polyp search and resection will be performed during the withdrawal phase in both groups. Insertion polypectomy will not be performed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 45 years or older undergoing colonoscopy for screening, surveillance, and positive FIT will be considered for enrollment.

Exclusion Criteria:

* familial adenomatous polyposis and hereditary non-polyposis CRC syndrome, personal history of CRC or inflammatory bowel disease, previous colonic resection, obstructive lesions of the colon, gastrointestinal bleeding, allergy to fentanyl, midazolam or propofol, American Society of Anesthesiology (ASA) classification of physical status grade 3 or higher, mental retardation, pregnancy, and refusal to provide a written informed consent.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiliang Cheng, MD, Principal Investigator — Evergreen General Hospital
Locations (1):
- Evergreen General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] le Clercq CM, Bouwens MW, Rondagh EJ, Bakker CM, Keulen ET, de Ridder RJ, Winkens B, Masclee AA, Sanduleanu S. Postcolonoscopy colorectal cancers are preventable: a population-based study. Gut. 2014 Jun;63(6):957-63. doi: 10.1136/gutjnl-2013-304880. Epub 2013 Jun 6. PMID 23744612
- [Background] Fuccio L, Frazzoni L, Hassan C, La Marca M, Paci V, Smania V, De Bortoli N, Bazzoli F, Repici A, Rex D, Cadoni S. Water exchange colonoscopy increases adenoma detection rate: a systematic review with network meta-analysis of randomized controlled studies. Gastrointest Endosc. 2018 Oct;88(4):589-597.e11. doi: 10.1016/j.gie.2018.06.028. Epub 2018 Jul 5. PMID 29981753
- [Background] Leung FW, Koo M, Cadoni S, Falt P, Hsieh YH, Amato A, Erriu M, Fojtik P, Gallittu P, Hu CT, Leung JW, Liggi M, Paggi S, Radaelli F, Rondonotti E, Smajstrla V, Tseng CW, Urban O. Water Exchange Produces Significantly Higher Adenoma Detection Rate Than Water Immersion: Pooled Data From 2 Multisite Randomized Controlled Trials. J Clin Gastroenterol. 2019 Mar;53(3):204-209. doi: 10.1097/MCG.0000000000001012. PMID 29505552
- [Background] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046
- [Derived] Cheng CL, Kuo YL, Hsieh YH, Tang JH, Leung FW. Comparison of Right Colon Adenoma Miss Rates Between Water Exchange and Carbon Dioxide Insufflation: A Prospective Randomized Controlled Trial. J Clin Gastroenterol. 2021 Nov-Dec 01;55(10):869-875. doi: 10.1097/MCG.0000000000001454. PMID 33074950

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Water Exchange (WE) Colonoscopy | CO2 Insufflation Colonoscopy
Started | 131 | 131
Completed | 131 | 131
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water Exchange (WE) Colonoscopy | CO2 Insufflation Colonoscopy | Total
Number analyzed (Participants) | 131 | 131 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (8.8) | 57.3 (8.3) | 57.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 64 | 134
  Male | 61 | 67 | 128
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 131 | 131 | 262

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adenomas and Hyperplastic Polyps Missed During Initial Right Colon Examination
Description: Lesions detected on the tandem (second) right colon examination are used for the calculation of adenoma and hyperplastic polyp miss rate. Right colon adenoma miss rate (AMR) and right colon hyperplastic polyp miss rate (HPMR) are calculated as the number of adenomas and hyperplastic polyps detected during the second right colon examination divided by the total number of adenoma and hyperplastic polyps detected during both the first and second right colon examinations.
Time Frame: One day
Measure: Mean (95% Confidence Interval); unit: percentage of all missed polyps
Arm/Group | Water Exchange (WE) Colonoscopy | CO2 Insufflation Colonoscopy
Number analyzed (Participants) | 131 | 131
percentage of all missed polyps | 18.0 [13.9 to 23.2] | 36.7 [30.0 to 44.8]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Water Exchange (WE) Colonoscopy | CO2 Insufflation Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/131
Other Adverse Events (participants affected / at risk) | 0/131 | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03845933/Prot_SAP_001.pdf